CLINICAL TRIAL: NCT02881827
Title: Biochemistry and Volumetric Analysis of Biofluid Salivary, Correlating the Flow, pH and Buffer Capacity With and Without Stimulation of the Masseter Muscle, Before and After Low-level Laser Irradiation
Brief Title: Saliva Analysis After Low-level Laser Therapy Application on the Masseter Muscle Located Above Parotid Salivary Gland
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Universidade do Vale do Paraíba (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: UNIVAP - Masulo 001
Record Dates: First submitted 2016-08-09; First posted 2016-08-29 (Estimated); Last update posted 2016-08-29 (Estimated); Status verified 2016-08

CONDITIONS: Saliva Altered
Keywords: Saliva; Low-level laser therapy; Masseter muscle; Salivary glands
MeSH Terms: interventions — Low-Level Light Therapy

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- Infrared Laser (Active Comparator): Using a laser in the infrared wave spectrum (780 nm)
  Interventions: Radiation: Low level laser therapy
- Red Laser (Active Comparator): Using laser red wave spectrum (662 nm)
  Interventions: Radiation: Low level laser therapy
- Placebo (Placebo Comparator): Simulation of treatment with the device switched off
  Interventions: Other: Placebo
- Control (Active Comparator): A scientific control group allows the experimental study of a variable at a time, and is a vital part of the scientific method. In a controlled experiment, two identical experiments are conducted. In one, the treatment - tested factor - is applied. In another - control - the tested factor is not applied
  For example, when testing a drug, it is important to carefully check the suspected drug effects are produced by the drug. Doctors can it with a double-blind study in a clinical trial: two ( statistically ) identical groups of patients are compared, one gets the drug and the other receives a placebo. Neither subjects nor investigators know which group receives the actual drug , which serves to prevent bias and isolating effects of such drugs.
  Interventions: Other: Control

INTERVENTIONS:
Radiation: Low level laser therapy — Supported by the physical phenomenon of stimulated emission postulated by Albert Einstein in 1916 the laser (light amplification by Stimulated Emission of Radiation) is a device consisting of solid source materials, liquid or gas that produces beams of light when excited by a source of energy. This bright feature is a particular type of electromagnetic radiation, which differs from that emitted by conventional incandescent sources. These are the effects attributable to LLLT analgesic, anti-inflammatory and biostimulates and has been widely used due to low power densities and wavelengths with a penetration capacity in tissues without the generation of photothermal effects, which makes its feasible use multiple applications in Health area.
  Arms: Infrared Laser; Red Laser
Other: Placebo — Simulation of treatment with the device switched off
  Arms: Placebo
Other: Control — A scientific control group allows the experimental study of a variable at a time, and is a vital part of the scientific method. In a controlled experiment, two identical experiments are conducted. In one, the treatment - tested factor - is applied. In another - control - the tested factor is not applied.
  For example, when testing a drug, it is important to carefully check the suspected drug effects are produced by the drug. Doctors can it with a double-blind study in a clinical trial: two (statistically) identical groups of patients are compared, one gets the drug and the other receives a placebo. Neither subjects nor investigators know which group receives the actual drug, which serves to prevent bias and isolating effects of such drugs.
  Arms: Control

SUMMARY:
The purpose of this study is to obtain experimental data on the possible changes that saliva may suffer when brought to low-level laser therapy protocols for analgesia in the masseter muscle, because this be on the Parotid salivary gland.

DETAILED DESCRIPTION:
Climate: The study will be conduced by Lasertherapy and Photobiology Center (CELAFO) at the Institute of Research and Development at the University of Vale do Paraíba (UNIVAP), which was air-conditioned with temperature at 22 ° C.

Volunteers: 30 male volunteers aged between 18 and 30 years.

Flow Analysis Salivary pH and saliva buffer capacity before LLLT and after LLLT: Two consecutive samples of whole saliva were obtained from each second volunteer. The first, unstimulated total saliva (UTS) and the second of stimulated total saliva (STS). Obtaining mechanically given by chewing a paraffin 5cm² fragment. The gathering was held in the afternoon and with the patient in breakfast for at least one hour. All the volunteers were instructed not to brush teeth or use mouthwash for one hour prior to saliva collection of the experiment. The samples were collected UTS and STS requesting voluntary saliva deposited directly into a sterile universal collector. Salivary samples were compared by the universal table salivary flow described by Saliva samples were centrifuged at 1200 rpm for 10 minutes. All saliva volume produced during the 5-minute period was measured using test tubes recorded in milliliters. The pH was measured by a pH meter device. To test the buffer capacity, the saliva (3 mL) was placed in a Falcon tube containing 9 mL of 0,005 normal hydrochloric acid, subjected to manual shaking for 10 seconds, then maintained at rest for 10 minutes with open Falcon tube, aiming evaporation gases such as carbon dioxide which could interfere with the analysis. After 10 minutes the pH was measured with litmus tape aid compared with the color scale provided by the manufacturer.

Low Level Laser Therapy (LLLT): The investigators used the LLLT after the first collection of saliva, control therapies were applied, placebo LLLT red and LLLT in the infrared.The treatment was applied with an interval of 7 days in a randomized, controlled, double-blind, by drawing lots. Irradiation of LLLT was conducted in eight (8) points on the skin in the masseter region. The distance between points was 1cm. To know exactly the location of points, transparency sheets were used (irradiation feedback) and reference points of each volunteer, as follows: point 1 commissure eyelid, point 2 in the tragus of the ear and point 3 on the labial commissure.The anticipated period of 15 minutes to occur the desired effects of LLLT was performed new material collection.

Data Analysis: The salivary flow data, pH and buffering capacity of saliva was analyzed using a analysis program statistics with the nonparametric Kruskal-Wallis test. The significance level was 5% (p <0.05)

ELIGIBILITY:
Inclusion criteria :

* Have all dental organs
* Male volunteers
* Age between 18 and 30 years
* Body mass index between 18.5 and 25 (normal) .

Exclusion Criteria:

Presence of problems that compromise the physiological activity of the masticatory system

* Neurological disorders
* Cerebral Palsy

parafunctions :

* Sucking fingers
* Nail biting
* Nibble objects
* Bruxism
* Mouth breathing .

Use of medication :

* Antihistamines
* Benzodiazepines
* Depressants of the central nervous system.

Temporomandibular dysfunction:

* Clenching of the teeth
* Bruxism
* Use of partial or full dentures .

Ages: 18 Years to 30 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 30 (Actual)
Dates: Start 2014-01; Primary Completion 2016-08 (Actual); Study Completion 2018-09 (Estimated)

PRIMARY OUTCOMES:
Increased salivary flow | 24 months
  Expect positive results of this research on the increased salivary flow , improved saliva buffer capacity as well as increased salivary pH enabling a better quality of life for patients.

SECONDARY OUTCOMES:
Improvement of the salivary pH | 24 months
  Expect positive results of this research on the increased salivary flow , improved saliva buffer capacity as well as increased salivary pH enabling a better quality of life for patients.

OTHER OUTCOMES:
Increase in saliva buffer capacity | 24 months
  Expect positive results of this research on the increased salivary flow , improved saliva buffer capacity as well as increased salivary pH enabling a better quality of life for patients.

CONTACTS AND LOCATIONS:
Locations (1):
- Leandro Júnio Masulo, São José dos Campos, São Paulo, Brazil

IPD SHARING:
Plan to Share IPD: Yes

REFERENCES:
- See also: Lattes Curriculum — http://lattes.cnpq.br/8398356986819265